CLINICAL TRIAL: NCT00639756
Title: Phase 2 Study to Determine if Allopurinol Blocks Features of Metabolic Syndrome Induced by Fructose Ingestion
Brief Title: The Effect of Allopurinol on Insulin Resistance and Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Mateo Orfila (Other)
Responsible Party: PEREZ-POZO, SANTOS E. LOPEZ-LILLO, JULIAN. JOHNSON, RICHARD, MATEO ORFILA HOSPITAL, University of Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IbSalut-M-001
Record Dates: First submitted 2008-03-10; First posted 2008-03-20 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Metabolic Syndrome
Keywords: Uric acid; Fructose; Hypertension; Insulin; Glucose; HOMA
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Insulin Resistance | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): Allopurinol given for 2 weeks with diet
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 300 mg
  Arms: 2
Drug: Placebo — Placebo given for 2 weeks
  Arms: 1

SUMMARY:
Studies in animals have found that allopurinol can markedly improve fructose induced metabolic syndrome. In this study we test the hypothesis that allopurinol may lower BP, reduce triglycerides, and improve metabolic parameters in subjects placed on a high fructose diet.

DETAILED DESCRIPTION:
60 male subjects, age 40 to 65 years of age, will be placed on a 3500kcal (55% carbohydrates containing 200 g fructose) for 2 weeks. Half will receive allopurinol mg/day (randomized). At the end of 2 weeks we measure a variety of parameters including fasting glucose and insulin levels (with calculation of HOMA index), serum lipids (including triglycerides and LDL/HDL cholesterol), sitting blood pressure, serum uric acid, weight, and various other measurements (C reactive protein, adiponectin and leptin levels, and urate redox products). Primary endpoint is insulin resistance. Secondary endpoints are blood pressure, lipids, uric acid, weight.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 40 -65 yrs

Exclusion Criteria:

* None

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (HOMA index) | 2 weeks
Blood pressure | 2 weeks
Triglycerides, HDL cholesterol | 2 weeks

SECONDARY OUTCOMES:
Adiponectin | 2 weeks
Leptin | 2 weeks
CRP level | 2 weeks
Weight gain | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Unit, Mateo Orfila Hospital, Menorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Johnson RJ, Perez-Pozo SE, Lillo JL, Grases F, Schold JD, Kuwabara M, Sato Y, Hernando AA, Garcia G, Jensen T, Rivard C, Sanchez-Lozada LG, Roncal C, Lanaspa MA. Fructose increases risk for kidney stones: potential role in metabolic syndrome and heat stress. BMC Nephrol. 2018 Nov 8;19(1):315. doi: 10.1186/s12882-018-1105-0. PMID 30409184
- [Derived] Perez-Pozo SE, Schold J, Nakagawa T, Sanchez-Lozada LG, Johnson RJ, Lillo JL. Excessive fructose intake induces the features of metabolic syndrome in healthy adult men: role of uric acid in the hypertensive response. Int J Obes (Lond). 2010 Mar;34(3):454-61. doi: 10.1038/ijo.2009.259. Epub 2009 Dec 22. PMID 20029377